CLINICAL TRIAL: NCT05885984
Title: Effects of Acceptance and Commitment Therapy on Fatigue Interference in Patients With Advanced Lung Cancer and Caregiver Burden: A Pilot Randomised Controlled Trial
Brief Title: Acceptance and Commitment Therapy on Fatigue Interference in Patients With Advanced Lung Cancer and Caregiver Burden (ACT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Association for contextual behavioral science (Unknown)
Responsible Party: Principal Investigator, Huiyuan LI, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CREC Ref. No. 2023.030
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer; Advanced Cancer; Caregiver Burden
Keywords: lung cancer; palliative care; Acceptance and Commitment Therapy; cancer-related fatigue; caregiver burden
MeSH Terms: conditions — Lung Neoplasms; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study. Participants in Group A receive Acceptance and Commitment Therapy in addition to health education. Participants in Group B receive health education.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor who is independent of the research will be trained before formally conducting data collecting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT group (Experimental): Participants in the intervention group will receive ACT intervention, consisting of six online sessions via video conferencing platform (The first two sessions for patient only, the third and fourth sessions for caregiver only, and the last two sessions for patient-caregiver dyads) of 60-90 min each (once/week), in addition to health education.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT) plus health education
- Health eduction control group (Other): Participants randomised to the health education control group will receive six weekly health education by a video-conferencing platform. The topics mainly include treatments and daily care during admission, medication instructions and side effects, diet and exercise advice, and retest recommendations when discharged.
  Interventions: Other: Health education

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) plus health education — Session 1: Reviewing experiences on struggles with CRF, realising consequence of controlling, introducing acceptance as an alternative, adopting virtual mindfulness. Education (patient): epidemiologic features of advanced lung cancer. Session 2: Separate thoughts/feelings related to CRF. Education (patient): treatments and symptoms of advanced lung cancer. Session 3: Reviewing caregiver's experiences of struggling with caregiving burden,introducing acceptance as an alternative. Education (caregiver): epidemiologic features of advanced lung cancer. Session 4: Separate caregivers' thoughts/feelings related to caregiving burden. Education (caregiver): treatments and symptoms of advanced lung cancer. Session 5:Understand the importance of values and clarifying personal values for dyads. Education (dyads): eating suggestions. Session 6: Emphasise ongoing value-based goals and commitment to actions for a meaningful cancer life for dyads. Education (dyads): exercising suggestions.
  Arms: ACT group
Other: Health education — Session 1: health education on the epidemiologic features of advanced lung cancer will be taught to patients. Session 2: health education on treatments and related symptoms of advanced lung cancer will be taught to patients. Session 3: health education on the epidemiologic features of advanced lung cancer will be taught to caregivers. Session 4: health education on treatments and related symptoms of advanced lung cancer will be taught to caregivers. Session 5: health education on eating suggestions for advanced lung cancer patients and caregivers will be taught. Session 6: health education on exercising suggestions for advanced lung cancer patients and caregivers will be taught.
  Arms: Health eduction control group

SUMMARY:
Lung cancer is a malignant tumour that has transformed from a single cancer disease into one of the most striking global health problems. Lung cancer has an insidious onset, and most patients are first diagnosed with the middle and advanced stages. Cancer-related fatigue is the most common and distressing symptom reported by lung cancer patients. For cancer patients, fatigue has a lasting impact on physical, psychological and social functions, and interferes with activities and participating in life events, thereby worsening the health-related quality of life. Family members have a key role in providing advanced lung cancer patients with informational, instrumental, and emotional support, which is crucial to patients' adaptation to the advanced illness and living a meaningful cancer life. Acceptance and Commitment Therapy (ACT) is the third-wave cognitive behavioural therapy to improve functioning and health-related quality of life by increasing psychological flexibility. The study aims to examine test the feasibility and acceptability, and preliminary effects of online ACT on fatigue interference in patients with advanced lung cancer and caregiver burden.

DETAILED DESCRIPTION:
A two-arm, assessor-blind randomised controlled trial will be conducted to investigate the effects of ACT on advanced lung cancer patients and caregivers compared to educational control. Participants in the same ward will be randomised at a 1:1 ratio to the intervention group or control group. Block randomization will be conducted by an independent research assistant using randomly varying block sizes of 4 and 6 to avoid selection bias. The study aims to examine the feasibility and acceptability, and preliminary effects of online ACT on fatigue interference in patients with advanced lung cancer and caregiver burden. The Specific objectives are:

1. To investigate the feasibility and acceptability of the online 6-week ACT in patients with advanced lung cancer and caregivers in rural areas in China;
2. To investigate the preliminary effects of the online 6-week ACT in patients with advanced lung cancer and caregivers in rural areas in China;
3. To explore how patients and caregivers perceive the ACT experience during the intervention process.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 or over;
2. diagnosed with stage III or stage IV lung cancer by pathological section or cytology;
3. lived in rural areas;
4. experienced unexplained fatigue syndrome: the score of 3 or more on the Fatigue Symptom Inventory (FSI);
5. able to provide informed consent and effectively collect data;
6. a consenting primary family caregiver; and
7. working phone service

Exclusion Criteria:

1. diagnosed with cognitive dysfunction or other mental illnesses that may interfere with their completion of treatment;
2. who are at critical condition; and
3. who are receiving or have just completed other lung cancer-related intervention programs within the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Eligibility rate | Before baseline
  The eligiblity rate is defined as the percentage of participants fulfilling the inclusion criteria amongst the participants screened for the eligibility
Recruimtment rate | Before baseline
  The recruitment rate is defined as the percentage of participants who consented to participate in the study amongst the participants eligible for the study
Attrition rate | After the 6-week intervention
  The attrition rate is defined as the percentage of participants who withdrew from the study before completion
Adherence rate | After the 6-week intervention
  The adherence rate is defined as the frequency of the practice of mindfulness and session attendance
Change from baseline in the score of fatigue interference assessed by The Fatigue Symptom Inventory at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 6-week intervention)
  A 13-item instrument that measures the intensity and interference of fatigue over the previous 7 days. The first four items are used to assess the intensity of fatigue, Item 5 - Item 11 are to assess the degree to which fatigue in the past week was judged to interfere with different aspects, such as general activity, bathe and dress ability, work activity, concentration ability, relation with others, enjoyment of life and mood, using a 11-point Likert scale ranging from 0 (no interference) to 10 (extreme interference). 0 indicates no fatigue and 127 indicates the worst fatigue intensity and interference.
Change from baseline in the score of caregiver burden assessed by The Zarit Caregiver Burden Inventory at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 6-week intervention)
  12 items score from 1(not always) to 5 (always) to assess caregiver burdens of caregivers of advanced lung cancer patients, including three domains: role strain, self-criticism, and negative emotion. The overall score can be obtained by adding all subscale scores. 12 indicates low caregiver burden and 60 indicates the highest caregiver burden.

SECONDARY OUTCOMES:
Change from baseline in the score of health-related quality of life assessed by Functional Assessment of Cancer Therapy - Lung, Version 4 at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 6-week intervention)
  36 items scored from 0 (not at all) to 4 (very much) to assess QoL of lung cancer patients, including 5 domains: physical, social/family, emotional, and functional well-being, and additional concerns about lung cancer. The overall score can be obtained by adding all subscale scores. 0 indicates no quality of life and 144 indicates the highest quality of life.
  Change= (One week after the intervention score - Baseline score)
Change from baseline in the score of meanfing of life assessed by The Meaning of Life questionnaire (MLQ) at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 6-week intervention)
  8 items score from 0 (not at all) to 7 (totall agree) to assess meaning of life of caregivers of advanced lung cancer patients, including 2 domains: the Presence of Meaning subscale and the Search for Meaning subscale. The overall score can be obtained by adding all subscale scores. 0 indicates no meaning of life and 56 indicates the highest meaning of life.
Change from baseline in the score of psychological flexibility assessed by Comprehensive assessment of Acceptance and Commitment Therapy processes at three months after the intervention | Baseline (T0) and post-intervention (T1, one week after the 6-week intervention)
  A comprehensive ACT process measure to evaluate the level of psychological flexibility (and constituent sub-process) within the ACT model with 18 items ranged from 18 to 90. 18 indicates low level of psychological flexibility and 90 indicates the high level of psychological flexibility.
Change from baseline in the score of mindful attention assessed by Mindful Attention Awareness Scale at one week after the intervention | Baseline (T0) and post-intervention (T1, one week after the 6-week intervention)
  The trait MAAS is a 15-item scale designed to assess a core characteristic of mindfulness, scored from 1 (almost never) to 6 (almost always). 15 indicates low level of awareness and attention to present moment and 90 indicates the high level of awareness and attention to the present moment.

OTHER OUTCOMES:
Acceptability of the intervention | After the 6-week intervention
  A convenience sample of 10 dyads in the intervention group will be recruited for focus group interviews to explore their ACT experience and overall satisfaction. The interview guide was developed based on the previous studies.

CONTACTS AND LOCATIONS:
Overall Officials: Cho Lee WONG, PhD, Study Director — The Nethersole School of Nursing, Chinese University of Hong Kong; Huiyuan LI, PhD, Principal Investigator — The Nethersole School of Nursing, Chinese University of Hong Kong
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Wong CL, Jin X, Wang N, Shi Z. Effects of acceptance and commitment therapy on fatigue interference in patients with advanced lung cancer and caregiving burden: protocol for a pilot randomised controlled trial. BMJ Open. 2024 Jul 23;14(7):e082090. doi: 10.1136/bmjopen-2023-082090. PMID 39043593